CLINICAL TRIAL: NCT01100736
Title: Characterisation of the Role of ETA and ETB Receptors in Regulating Plasma ET-1 and the Vasodilator Response to ET-3 in Man
Brief Title: Role of Endothelin-A (ETA) and Endothelin-B (ETB) Receptors in the Vasodilatory Response to Endothelin-3 (ET-3)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Encysive Pharmaceuticals (Industry)
Responsible Party: Professor David Webb, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2008/W/CRC/01; 08/S1102/1
Record Dates: First submitted 2010-03-30; First posted 2010-04-09 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Arterial Hypertension; Vasodilation; Vasoconstriction
Keywords: Forearm Blood Flow; Vasodilation; Vasoconstriction; Endothelin System; Endothelin-1; Endothelin-3; Endothelin antagonists; Bosentan; Sitaxsentan; Endothelin; Regional Blood Flow
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Aneurysm | interventions — Bosentan; sitaxsentan; Endothelin-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bosentan (Experimental): Bosentan 125mg twice daily will be taken for 7 days, before ET-1 plasma sample taken. ET-3 infusion (5mins) and associated forearm blood flow study (60 mins) will also occur after 7 days of bosentan therapy
  Interventions: Drug: Bosentan; Biological: Endothelin-3
- Sitaxsentan (Experimental): Sitaxsentan 100mg once daily + placebo tablet will be taken for 7 days, before ET-1 plasma sample taken. ET-3 infusion (5mins) and associated forearm blood flow study (60 mins) will also occur after 7 days of sitaxsentan therapy
  Interventions: Drug: Sitaxsentan; Drug: Placebo; Biological: Endothelin-3
- Placebo (Placebo Comparator): Placebo tablet twice daily will be taken for 7 days, before ET-1 plasma sample taken. ET-3 infusion (5mins) and associated forearm blood flow study (60 mins) will also occur after 7 days of placebo therapy
  Interventions: Drug: Placebo; Biological: Endothelin-3

INTERVENTIONS:
Drug: Bosentan — Bosentan 125mg tablets, orally, twice daily for 7 days
  Other Names: Tracleer
  Arms: Bosentan
Drug: Sitaxsentan — Sitaxsentan 100mg tablets, orally, once daily for 7 days
  Other Names: Thelin
  Arms: Sitaxsentan
Drug: Placebo — Placebo tablets taken twice daily, orally, for 7 days (placebo arm) or once daily for 7 days (sitaxsentan arm)
  Arms: Placebo; Sitaxsentan
Biological: Endothelin-3 — 5 minute local intra-arterial infusion of endothelin-3 at a rate of rate of 60 pmol/min, during forearm blood flow studies

SUMMARY:
Endothelin-1 (ET-1) has been linked to a number of conditions including pulmonary arterial hypertension (PAH). ET-1 acts via 2 receptors, ETA and ETB. The ET-1 receptor blockers bosentan and sitaxsentan have been shown to be beneficial in patients with PAH. Bosentan blocks both ETA and ETB receptors. Sitaxsentan selectively blocks ETA receptors. Theoretically, selective ETA blockade may be associated with greater vasodilation and clearance of ET-1 by leaving the ETB receptor unblocked. This has not been directly studied in humans.

We aim to investigate the endothelial ETB-mediated vascular responses between bosentan and sitaxsentan by using a ETB selective agonist (ET-3). We hypothesise that at clinically relevant doses:

* Bosentan will show evidence of ETB receptor blockade compared to sitaxsentan and placebo.
* These effects will be confirmed by 2 functional markers of ETB receptor antagonism: plasma ET-1 (a very sensitive, but not necessarily clinically relevant marker), and the forearm vasodilator response to ET-3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and post-menopausal women
* Age 18-70 years
* BMI 18-35 kg/m2

Exclusion Criteria:

* Are mentally or legally incapacitated
* Have donated blood within the last 4 weeks
* Have a history of past or present drug or alcohol abuse
* Have participated in another clinical trial within 1 month
* Are considered to be at a high risk of HIV or Hepatitis B
* Are taking routine medicines
* Are women taking hormone replacement therapy
* Have significant medical or psychiatric illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Plasma ET-1 after 7-day administration of bosentan, sitaxsentan and placebo | 7 days
Responses to ET-3 (maximum vasodilation after ET-3 administration and area under the curve of vasodilation) after bosentan compared with the results from sitaxsentan and placebo. | 60 mins

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Western General Hospital, Edinburgh, Scotland, United Kingdom